CLINICAL TRIAL: NCT02164643
Title: Longitudinal Study of Brain Amyloid imaGing in MEMENTO
Acronym: MEMENTOAmyGing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Fondation Plan Alzheimer (Other); GE Healthcare (Industry); Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2010/47 A
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Alzheimer's Disease (AD) and Related Disorders
Keywords: Alzheimer's disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — flutemetamol; florbetapir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Florbetapir (18F) (Experimental)
  Interventions: Drug: Florbetapir (18F)
- Flutemetamol (18F) (Experimental)
  Interventions: Drug: Flutemetamol (18F)

INTERVENTIONS:
Drug: Flutemetamol (18F)
  Arms: Flutemetamol (18F)
Drug: Florbetapir (18F)
  Arms: Florbetapir (18F)

SUMMARY:
A Multicenter national longitudinal cohort study including at least 800 individuals consecutively recruited from French Research Memory Centers and followed-up over 24 month and included in Memento.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia in the elderly, affecting approximately 7.3 million people in Europe. AD is a clinicopathologic entity for which the definitive diagnosis requires both the presence of the clinical signs of dementia and pathological evidence of amyloid plaque in the brain (obtained at autopsy).

Currently, diagnosis of AD at early stage of the disease is hampered by the lack of noninvasive and validated biomarkers of the underlying pathology. On one hand, it is suggested that between 10% and 20% of patients currently diagnosed with AD, based on clinical evidence solely, lack AD pathology at autopsy, and on the other hand community physicians may not diagnose AD in 33% of patients with mild signs and symptoms. Thus, there is a need for validated diagnostic biomarker that could help clinicians separate patients who do not have AD from those who have pathological signs and should be referred for further evaluation and care management. Furthermore, little is known on the prognosis value for dementia conversion of current biomarkers of AD pathology at a preclinical or presymptomatic stage.

Recently, 18F-labeled positron emission tomography (PET) imaging agents have been developed that bind with high affinity to the amyloid-β (Aβ) peptide fibrils that constitute amyloid plaques, and thus, have potential value as an imaging biomarkers for amyloid deposits in subjects with cognitive impairment or isolated cognitive complaints.

The principal objective of this ancillary study is to investigate the prospective association between PET amyloid load, measured twice two years apart, through either Florbetapir (18F) or Flutemetamol (18F) radioligands, and dementia incidence over up to 5 years of follow-up in a sample of individuals presenting with a spectrum of cognitive profiles ranging from isolated cognitive complaints to cognitive deficits without dementia.

The secondary objectives are the following:

* To assess the association between change in amyloid load and clinical evolution of participants (both functional and cognitive)
* To estimate the prevalence of new research criteria for preclinical Alzheimer's disease
* To investigate long-term outcome of preclinical Alzheimer's disease according to NIA-AA criteria
* To assess the determinants of change in amyloid load over two years
* To study the interrelationships between biomarkers
* To assess the added value of amyloid binding agent (Florbetapir (18F) and Flutemetamol (18F)) in combination with other biomarkers (neuropsychological, genetics, plasma, serum, CSF, structural neuroimaging, 18F-FDG-PET) to predict clinical dementia onset
* To assess the diagnostic accuracy of amyloid agent Florbetapir (18F) and Flutemetamol (18F) to differentiate AD from other types of dementia (differential diagnosis)
* To study the link between amyloid binding agent and survivalstudy design

ELIGIBILITY:
Inclusion Criteria:

* To be included in MEMENTO
* To have signed a specific MEMENTO-AmyGing informed consent form, prior to any amyloid PET procedures
* To have had or agreed to have 18F-FDG PET scan in MEMENTO
* To tolerate the (18F) PET scan procedures, in the opinion of the clinical site investigator
* Clinical Dementia Rating scale <0.5 and not demented

Exclusion Criteria:

* To have a current clinically significant psychiatric condition that neurologists/geriatricians feel would preclude the ability to have a research PET scan
* To be pregnant or breastfeading women
* To have Hypersensitivity to the tracer or to the excipient listed in the summary of the product carateristics (florbetapir Amyvid®) or the Investigator's Brochure (flutemetamol)
* To have a relevant history of severe drug allergy or hypersensitivity (relevant severe drug allergies should be determined by the clinical site investigator or co-clinical site investigator). If a subject has a history of severe drug allergies, it may be dangerous for them to participate in a study with a novel compound
* To have ever participated in an experimental study with an amyloid targeting agent (e.g. anti-amyloid immunotherapy, γ-secretase or γ-secretase inhibitor) unless it can be documented that the subject received only placebo during the course of the trial
* To receive any investigational medications, or have participated in a trial with investigational medications within the last 30 days
* To have participated less than 1 year ago in a biomedical research with injection of one of the amyloid radioligand or to be enrolled in an ongoing biomedical research including amyloid PET scan
* To have had a radiopharmaceutical imaging or treatment procedure within 7 days prior to the study imaging session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2014-06-10 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Progression to clinical dementia stage according to standardized classifications (DSM-IV and NINCDS-ADRDA) as described in the MEMENTO protocol. | 24 months from baseline

SECONDARY OUTCOMES:
Longitudinal evolution of amyloid load measured through either Florbetapir (18F) or Flutemetamol (18F) | 24 months from baseline
Speed of cognitive decline based on change in cognitive performances | 24 months from baseline
Longitudinal evolution of biomarkers measured from blood, CSF, structural neuroimaging (MRI) and glucose metabolism molecular neuroimaging (18F-FDG PET). | 24 months from baseline
Mortality | 24 months from baseline
Loss of autonomy based on functional activity assessment | 24 months from baseline
Institutionalization | 24 months from baseline
Cardiovascular event (Stroke and Coronary events) | 24 months from baseline
Quality of life | 24 months from baseline
Prodromal AD (Pre-symptomatic dementia) | 24 months from the baseline
Etiology of dementia, when converted | 24 months from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve CHENE, Prof, Principal Investigator — CIC-EC7 - ISPED - CHU de Bodeaux; Geneviève CHENE, Prof, Study Chair — CIC-EC7 - ISPED - CHU de Bordeaux; Carole DUFOUIL, Director, Study Director — CIC-EC7 - ISPED - CHU de Bordeaux; Florence PASQUIER, Prof, Study Director — Head of Lille Memory Clinic, CHRU Lille; Marie-Odile HABERT, Prof, Study Director — Head of Molecular Imaging Work package for the Center for Image Acquisition and Processing - CHU Pitié-Salpêtrière, AP-HP
Locations (26):
- France (26):
  - CHU d'Angers, Angers
  - CHU de Besançon, Besançon
  - AP-HP - Avicenne, Bobigny
  - CHU de Bordeaux - Pellegrin, Bordeaux
  - CHU de Bordeaux - Hôpital Xavier-Arnozan, Bordeaux
  - CHU de Brest, Brest
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - Hospices civils de Lyon, Lyon
  - AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nice, Nice
  - AP-HP - Hôpital BROCA, Paris
  - AP-HP - Hôpital LARIBOISIERE, Paris
  - Ap-Hp La Pitié-Salpêtrière, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Rouen, Rouen
  - CHU de Saint-Etienne - Hôpital de la charité, Saint-Etienne
  - CHU de Saint-Etienne - Hôpital Nord, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse - Hôpital Purpan, Toulouse
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours

REFERENCES:
- [Derived] Ackley S, Calmasini C, Bouteloup V, Hill-Jarrett TG, Swinnerton KN, Chene G, Dufouil C, Glymour MM; MEMENTO Cohort Study Group and DPUK. Contribution of Global Amyloid-PET Imaging for Predicting Future Cognition in the MEMENTO Cohort. Neurology. 2024 Mar 26;102(6):e208054. doi: 10.1212/WNL.0000000000208054. Epub 2024 Feb 27. PMID 38412412